CLINICAL TRIAL: NCT01961167
Title: Evaluation of the GORE® VIABAHN® BALLOON EXPANDABLE ENDOPROSTHESIS (VIABAHN BX) for the Treatment of Occlusive Disease in the Common and External Iliac Arteries
Brief Title: Evaluation of the GORE® VIABAHN® BALLOON EXPANDABLE ENDOPROSTHESIS (VIABAHN BX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBX 13-05
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Common Iliac Artery Occlusive Disease; External Iliac Artery Occlusive Disease; Peripheral Arterial Disease
Keywords: PAD; Stent; Claudication; VIABAHN; Gore; Endoprosthesis; Vascular Diseases; Cardiovascular Diseases; Iliac Occlusive Disease; Balloon Expandable; Stent Graft; VBX
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gore VIABAHN BX (Experimental): Balloon expandable stenting of iliac occlusive disease
  Interventions: Device: Stenting of common and/or external iliacs

INTERVENTIONS:
Device: Stenting of common and/or external iliacs — Balloon expandable stenting of iliac occlusive disease

SUMMARY:
The primary objective of the VBX13-05 clinical study is to evaluate the safety and efficacy of VIABAHN BX for the treatment of arterial occlusive disease in patients with de novo or restenotic lesions in the common and/or external iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old;
* Patient is male, infertile female, or female of childbearing potential practicing an acceptable method of preventing pregnancy;
* Patient or legal representative is willing to give written informed consent;
* Patient is capable of complying with protocol requirements, including all follow-up visits;
* Patient has symptomatic claudication or rest pain without tissue loss (Rutherford Categories 2-4).
* Patient has de novo or restenotic target lesion(s) in the common and/or external iliac artery

Exclusion Criteria:

* Patient has a life expectancy of less than 1 year;
* Patient has a known allergy to stent graft components, including stainless steel or heparin;
* Patient has a known intolerance to antiplatelet, anticoagulant, or thrombolytic medications that would prevent compliance with the protocol;
* Patient has a condition (unrelated to the study) that is expected to require indefinite, or lifelong, anticoagulation
* Patient has had vascular access / catheterization in the lower extremity within 30 days of study enrollment;
* Patient has had a previous or planned coronary intervention within 30 days prior to enrollment in this study or required at time of study procedure; Patient has had a previous or planned bypass surgery in the target leg, or a bypass that occurs at the time of the study procedure;
* Patient is currently participating in this or another investigative clinical study.
* Patient has evidence of angiographically visible thrombus within or adjacent to the target lesion(s);
* Patient has aneurysmal dilation proximal or distal to the target lesion(s) that would interfere with the placement of the device;
* Patient has a target lesion requiring atherectomy or any ablative device to facilitate stent delivery;
* Patient has a target lesion situated in such a way that an implanted device will prevent blood flow or perfusion to the internal iliac artery if patent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MB ChB, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gore VIABAHN BX
Started | 27
Completed (Completion of primary endpoint milestone at 30 days and secondary endpoints at 6 months.) | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects meeting all eligibility criteria.
Groups:
- Iliac Stenting: Balloon expandable stenting of iliac occlusive disease
  Stenting of common and/or external iliacs: Balloon expandable stenting of iliac occlusive disease
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 27

OUTCOME MEASURES:

1. Primary Outcome: Composite of Major Adverse Events (MAEs)
Description: Percentage of study subjects experiencing a major adverse event (MAE) defined as:
  * Device- or procedure-related death within 30 days of the index procedure; and
  * Myocardial Infarction (MI) occurring within 30 days of the index procedure; and
  * Amputation above the metatarsals in the treated leg, resulting from a vascular event, occurring within 30 days of the index procedure.
Time Frame: 30 days
Population: Population includes enrolled subjects who either experienced the defined event or were followed for at least 30 days.
Measure: Number (95% Confidence Interval); unit: percentage of subjects experiencing MAE
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of subjects experiencing MAE | 0 [0 to 12.8]

2. Secondary Outcome: Acute Procedural Success
Description: Number of subjects who experience acute procedural success defined as less than or equal to 30% residual stenosis prior to procedure completion and no device- or procedure-related SAEs before discharge at day 1.
Time Frame: Discharge
Population: Population includes subjects followed through discharge at day 1 and had relevant procedural data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 27

3. Secondary Outcome: Thirty-day Clinical Success
Description: Number of subjects who experienced 30-day clinical success defined as an improvement of at least one Rutherford Category at the 30-day visit as compared to pre-procedure and no device- or procedure-related serious adverse events (SAEs) within 30 days of the index procedure.
  Rutherford categories include:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 25

4. Secondary Outcome: Primary Patency
Description: Kaplan-Meier estimate of primary patency at 30 days. Primary patency is defined as blood flow in the treated segment(s), without reintervention.
Time Frame: 30 Days
Population: Analysis includes subjects followed for at least 30 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

5. Secondary Outcome: Primary Patency
Description: Kaplan-Meier estimate of primary patency at 6 months. Primary patency is defined as blood flow in the treated segment(s), without reintervention.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 180 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

6. Secondary Outcome: Primary Assisted Patency
Description: Kaplan-Meier estimate of primary assisted patency at 30 days. Primary assisted patency is defined as blood flow maintained with or without reintervention in the originally treated segment(s), including the proximal and distal margins.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

7. Secondary Outcome: Primary Assisted Patency
Description: Kaplan-Meier estimate of primary assisted patency at 6 Months. Primary assisted patency is defined as blood flow maintained with or without reintervention in the originally treated segment(s), including the proximal and distal margins.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 180 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: Lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Lesions | 100 [100 to 100]

8. Secondary Outcome: Secondary Patency
Description: Kaplan-Meier estimate of secondary patency at 30 days. Secondary patency is defined as presence of blood flow, with or without reintervention, in the originally treated segment(s), including the proximal and distal margins.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

9. Secondary Outcome: Secondary Patency
Description: Kaplan-Meier estimate of secondary patency at 6 months. Secondary patency is defined as presence of blood flow, with or without reintervention, in the originally treated segment(s), including the proximal and distal margins.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 180 days and had relevant data.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

10. Secondary Outcome: Freedom From Target Lesion(s) Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 30 days. TLR is defined as revascularization occurring within the treated segment(s) by means of a percutaneous vascular intervention, surgical bypass, thrombolysis, or other invasive means.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

11. Secondary Outcome: Freedom From Target Lesion(s) Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 6 months. TLR is defined as revascularization occurring within the treated segment(s) by means of a percutaneous vascular intervention, surgical bypass, thrombolysis, or other invasive means.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 180 days.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of lesions | 100 [100 to 100]

12. Secondary Outcome: Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 30 days. TVR is defined as revascularization of the vessel treated at the time of the index procedure by means of a percutaneous vascular intervention, surgical bypass, thrombolysis, or other invasive means.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Number (95% Confidence Interval); unit: Vessel
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Vessel | 100 [100 to 100]

13. Secondary Outcome: Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 6 months. TVR is defined as revascularization of the vessel treated at the time of the index procedure by means of a percutaneous vascular intervention, surgical bypass, thrombolysis, or other invasive means.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 180 days.
Measure: Number (95% Confidence Interval); unit: percentage of vessel
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
percentage of vessel | 100 [100 to 100]

14. Secondary Outcome: Number of Participants With a Change in Rutherford Category
Description: Change in Rutherford Category from pre-procedure at 30 days.
  Rutherford categories include:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 30 Days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants
  Improved | 25
  Maintained | 1
  Worsened | 1

15. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Change in Rutherford Category from pre-procedure at 6 months.
  Rutherford categories include:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 22
Participants
  Improved | 19
  Maintained | 1
  Worsended | 2

16. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: Change in Ankle Brachial Index (ABI) from pre-procedure at 30 days. Larger values indicate a better outcome. The ABI is the systolic pressure at the ankle, divided by the systolic pressure at the arm
Time Frame: 30 Days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Mean (Full Range); unit: ratio
Units Other Than Participants: limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Number analyzed (limbs) | 39
ratio | .15 [-0.16 to 0.53]

17. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: Change in Ankle Brachial Index(ABI) from pre-procedure at 6 months. Larger values indicate a better outcome.The ABI is the systolic pressure at the ankle, divided by the systolic pressure at the arm
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Mean (Full Range); unit: ratio
Units Other Than Participants: limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Number analyzed (limbs) | 33
ratio | .15 [-0.17 to 0.69]

18. Secondary Outcome: Freedom From Major Adverse Events (MAEs)
Description: Number of subjects experiencing freedom from procedure- or device-related events causing death, occurring within 30 days of the index procedure; and myocardial infarction (MI) occurring within 30 days of the index procedure; and target lesion revascularization (TLR) occurring within 6 months of the index procedure; and major amputation of the treated leg(s), resulting from a vascular event, occurring within 6 months of the index procedure.
Time Frame: 6 months
Population: Population includes number of subjects enrolled into the study who either had defined event or were followed for at least 150 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 27

19. Secondary Outcome: Change in Functional Status - EQ5D- Mobility
Description: Change in functional status (EQ5D - Mobility) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants
  Improved | 12
  Maintained | 12
  Worsened | 2

20. Secondary Outcome: Change in Functional Status - EQ5D- Mobility
Description: Change in functional status (EQ5D - Mobility) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Patient population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants
  Improved | 10
  Maintained | 10
  Worsened | 3

21. Secondary Outcome: Change in Functional Status - EQ5D - Self Care
Description: Change in functional status (EQ5D - Self Care) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants
  Improved | 0
  Maintained | 26
  Worsened | 0

22. Secondary Outcome: Change in Functional Status - EQ5D - Self Care
Description: Change in functional status (EQ5D - Self Care) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants
  Improved | 0
  Maintained | 22
  Worsened | 1

23. Secondary Outcome: Change in Functional Status - EQ5D - Usual Activities
Description: Change in functional status (EQ5D - Usual Activities) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants
  Improved | 13
  Maintained | 12
  Worsened | 1

24. Secondary Outcome: Change in Functional Status - EQ5D - Usual Activities
Description: Change in functional status (EQ5D - Usual Activities) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants
  Improved | 8
  Maintained | 14
  Worsened | 1

25. Secondary Outcome: Change in Functional Status - EQ5D - Pain/Discomfort
Description: Change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants
  Improved | 14
  Maintained | 10
  Worsened | 2

26. Secondary Outcome: Change in Functional Status - EQ5D - Pain/Discomfort
Description: Change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants
  Improved | 10
  Maintained | 12
  Worsened | 1

27. Secondary Outcome: Change in Functional Status - EQ5D - Anxiety/Depression
Description: Change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants
  Improved | 5
  Maintained | 20
  Worsened | 1

28. Secondary Outcome: Change in Functional Status - EQ5D - Anxiety/Depression
Description: Change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants
  Improved | 2
  Maintained | 21
  Worsened | 0

29. Secondary Outcome: Change in Functional Status - EQ5D- Own Health State
Description: Change in functional status (EQ5D - Own Health State) from pre-procedure at 30 days. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 25
Participants
  Improved | 4
  Maintained | 19
  Worsened | 2

30. Secondary Outcome: Change in Functional Status - EQ5D- Own Health State
Description: Change in functional status (EQ5D - Own Health State) from pre-procedure at 6 months. EQ5D is a standard instrument for use as a measure of health outcome.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 22
Participants
  Improved | 3
  Maintained | 17
  Worsened | 2

31. Secondary Outcome: Number of Participants With Improvement in Differential Diagnoses at 30 Days - Walking Impairment Questionnaire (WIQ)
Description: Patient reported outcome based on study questionnaire. Percentage of subjects with improvement on WIQ from pre-procedure at 30 days.
Time Frame: 30 day
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 26
Participants | 20

32. Secondary Outcome: Number of Participants With Improvement in Differential Diagnoses at 180 Days - Walking Impairment Questionnaire (WIQ)
Description: Patient reported outcome based on study questionnaire. Percentage of subjects with improvement on WIQ from pre-procedure at 180 days.
Time Frame: 6 Months
Population: Population includes subjects followed for at least 6 Months and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 23
Participants | 17

33. Other Pre Specified Outcome: Device or Procedure-related Death
Description: Number of subjects experiencing a device or procedure-related death within 30 days - component of primary outcome.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 0

34. Other Pre Specified Outcome: Freedom From Myocardial Infarction (MI)
Description: Number of subjects experiencing a myocardial infarction (MI) within 30 days - component of primary outcome.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 0

35. Other Pre Specified Outcome: Freedom From Major Amputation of the Treated Leg(s)
Description: Number of subjects experiencing a major amputation of the treated leg(s), resulting from a vascular event within 6 months - component
Time Frame: 6 Months
Population: Population includes subjects followed for at least 150 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 27
Participants | 0

ADVERSE EVENTS:
Time Frame: Through 6 months
Arm/Group | Iliac Stenting
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliac Stenting (N=27)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No